CLINICAL TRIAL: NCT03603548
Title: Comparison of Safety and Efficacy of Two Variants of Prolonged - Released Tacrolimus (Advagraf vs. Envarsus ) in Patients After Liver Transplantation : Single Center Randomised Control Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WarsawMUAdvEnv
Record Dates: First submitted 2018-07-19; First posted 2018-07-27 (Actual); Last update posted 2018-07-27 (Actual); Status verified 2018-07

CONDITIONS: Liver Transplant Rejection; Immunosuppression
MeSH Terms: interventions — Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Advagraf (Active Comparator)
  Interventions: Drug: Advagraf
- Envarsus (Experimental)
  Interventions: Drug: Envarsus

INTERVENTIONS:
Drug: Envarsus — Patients after liver transplantation initially treated with traditional Tacrolimus variant- Prograf, switched on day 10 after OLTx on prolonged released Tacrolimus variant in 1:1 ratio ( Advagraf vs. Envarsus)
  Arms: Envarsus
Drug: Advagraf — Patients after liver transplantation initially treated with traditional Tacrolimus variant- Prograf, switched on day 10 after OLTx on prolonged released Tacrolimus variant in 1:1 ratio ( Advagraf vs. Envarsus)
  Arms: Advagraf

SUMMARY:
Adult patients after liver transplantation initially treated with traditional Tacrolimus variant- Prograf, switched on day 10 after orthotropic liver transplantation (OLTx) on prolonged released Tacrolimus variant in 1:1 ratio ( Advagraf vs. Envarsus)

ELIGIBILITY:
Inclusion Criteria:

adults 18- 70 after liver transplantation due to liver cirrhosis primary liver transplantation

Exclusion Criteria:

liver transplantation due to liver cirrhosis and hepatocellular carcinoma (HCC) retransplantation renal impairment Parkinson disease

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2018-07-09 (Actual); Primary Completion 2023-07-09 (Estimated); Study Completion 2023-07-09 (Estimated)

PRIMARY OUTCOMES:
acute rejection | 12 months
chronic rejection | 5 years
tremor | 12 months
de novo diabetes | 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Warsaw Medical University, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: Undecided